CLINICAL TRIAL: NCT04805996
Title: The eHealth Diabetes Remission Trial - Pilot Study
Acronym: eDIT-pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Julia Otten (Other)
Collaborators: Region Västerbotten (Other Government)
Responsible Party: Sponsor-Investigator, Julia Otten, MD, PhD, Umeå University
Organization: Umeå University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 2021-00318
Record Dates: First submitted 2021-03-13; First posted 2021-03-18 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Type 2 Diabetes
Keywords: diabetes remission; weight loss; low-calorie diet; eHealth
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diabetes remission using total diet replacement and eHealth contact with the healthcare provider (Experimental): This study has only one arm and no comparator.
  Interventions: Behavioral: Diabetes remission using total diet replacement and eHealth contact with the healthcare provider

INTERVENTIONS:
Behavioral: Diabetes remission using total diet replacement and eHealth contact with the healthcare provider — Participants will replace usual foods with the commercially available total diet replacement Modifast (Impolin AB), which is delivered to them during the study period without any cost. Participants will be supplied with a scale, a finger-stick blood glucose meter and a blood pressure monitor and will be advised to measure body weight, fasting blood glucose and blood pressure every morning. The results are registered in the mobile phone application Telia Health Monitoring (Telia Sweden AB) and are wirelessly transmitted to the study team.

SUMMARY:
Ten study participants will consume a low-calorie total diet replacement for 12 weeks, have a 6-week food reintroduction phase (week 13-18) and continue with the weight loss maintenance phase until the end of the study (week 19-26). The weight loss goal is 15 kg (or 15% if body weight is bellow 80 kg). The primary study outcome iw weight loss after 6 months and the co-primary outcome is diabetes remission after 6 months (HbA1c < 48 mmol/mol). During the weight maintenance phase, if weight regain occurs or if HbA1c increases a rescue plan of total diet replacement will be recommended.

The participants will be supplied with the total diet replacement Modifast free of charge. Participants will be supplied with a scale, a finger-stick blood glucose meter and a blood pressure monitor. Participants will be advised to measure body weight, blood glucose and blood pressure every morning. The results are registered in the mobile phone application Telia Health Monitoring and are wirelessly transmitted to the project's physician, nurse and dietician. At the beginning of the food reintroduction phase the participants will receive an activity tracer and will be advised to increase their physical activity. Primary and secondary outcome measures will be estimated at the beginning and after 3 and 6 months. At the end of the study, all participants will take part in an individual semi-structured interview to investigate the participants' experience of diabetes remission and of the eHealth contact with the healthcare provider. After participants have completed the study, they will be followed at least once per year by obtaining data on blood sugar, HbA1c, body weight, blood pressure, medication usage and diabetes complications from the healthcare computer system.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes with diabetes duration 0 to 6 years
* BMI 27-45 kg/m2
* Owning a smartphone
* HbA1c 43-107 mmol/mol during the past 12 months (48-107 mmol/mol without blood sugar lowering medication)

Exclusion Criteria:

* Insulin treatment
* Weight loss 5 kg or more during the past 6 months
* Treatment with weight loss medication
* Diagnosed eating disorder
* eGFR < 30 ml/min/1.73m2
* Substance abuse
* Cancer
* Myocardial infarction during the past 6 months
* Severe heart failure
* Pregnancy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-23 (Actual); Primary Completion 2022-01-29 (Actual); Study Completion 2022-01-29 (Actual)

PRIMARY OUTCOMES:
Weight loss | 6 months
  Weight loss goal of 15 kg, measured at the research facilities
HbA1c | 6 months
  The goal is diabetes remission with HbA1c < 48 mmol/mol without any diabetes medication. (Secondary goal < 42 mmol/mol.)

SECONDARY OUTCOMES:
Semi-structured interviews | 6 months
Fasting blood glucose | Daily measurements up to 6 months
  Partial diabetes remission (< 7.0 mol/l), complete diabetes remission (<6.1 mol/l)
Fasting blood glucose | 6 months
  Partial diabetes remission (<7.0 mol/l), complete diabetes remission (<6.1 mol/l) without diabetes medication.
P-glucose 120 minutes after the oral glucose tolerance test | 6 months
  Measured at the research facilities
Insulin secretion | At baseline, 3 months and 6 months
  Measured with oral glucose tolerance test
Insulin sensitivity | At baseline, 3 months and 6 months
  Measured with oral glucose tolerance test
Metabolic flexibility | At baseline, 3 months and 6 months
  Measured with indirect calorimetry during oral glucose tolerance test
Blood pressure (systolic/diastolic) | At baseline, 3 months and 6 months
  Measured at the research facilities
Blood pressure (systolic/diastolic) | Daily measurements up to 6 months
  Measured at home
Blood pressure medication | 6 months
  Change of blood pressure medication during the study
Body weight | Daily measurements up to 6 months
  Measured at home
HbA1c | Monthly measurement up to 6 months
  Measured at home
Diabetes medication | 6 months
  Change of diabetes medication during study duration
Plasma lipid profile | At baseline, 3 months and 6 months
  Measured at the research facilities
Waist circumference | Baseline, 3 months and 6 months
  Measured in cm at the research facilities
EQ-5D-5L | At baseline, 3 months and 6 months
  Questionnaire
Food frequency form | At baseline and 6 months
  Questionnaire
Daily steps | During the second three months of the study
  Measured with activity tracker
HbA1c follow up | Yearly up to 20 years
  Collected from patient journals after study completion
Body weight follow up | Yearly up to 20 years
  Collected from patient journals after study completion
Blood pressure follow up (systolic/diastolic) | Yearly up to 20 years
  Collected from patient journals after study completion
Antidiabetic medication usage follow up | Yearly up to 20 years
  Collected from patient journals after study completion
Blood pressure medication usage follow up | Yearly up to 20 years
  Collected from patient journals after study completion
Diabetes complications follow up | Yearly up to 20 years
  Collected from patient journals and registries after study completion

CONTACTS AND LOCATIONS:
Overall Officials: Julia Otten, MD, PhD, Principal Investigator — Umeå University
Locations (1):
- Department of Public Health and Clinical Medicine, Medicine, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No